CLINICAL TRIAL: NCT05966103
Title: The Effects of Scapulothoracic Exercises on Postural Stability, Muscle Strength, Muscular Endurance and Proprioception in Sedentary Individuals With Cranio-Servico-Mandibular Malalignment
Brief Title: Efficacy of Scapulothoracic Exercises on Postural Stability, Proprioception, Muscular Features and Mandibular Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Collaborators: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0232
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Forward Head Posture
Keywords: Musculoskeletal Rehabilitation; Temporomandibular Joint Treatment; Scapulothoracic Exercises; Cranio-Cervico-Mandibular Malalignment
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Comparative Double-Blind Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Evaluations were done by a different physical therapist. The physiotherapist who administered the treatment was different. In addition, the participants did not know which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Exercise Group (Control Group) (Active Comparator): Conventional neck exercises were applied to the control group.
  Interventions: Other: Exercises
- Scapulothoracic Exercise (Treatment Group) (Experimental): In the treatment group, scapulothoracic exercises were applied in addition to conventional neck exercises.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — For control group; Cervical conventional exercises. For treatment group; scapulothoracic exercises including strengthening, proprioceptive and stabilization exercises in addition to cervical conventional exercises

SUMMARY:
The goal of this Randomized, Double-Blind, Clinical Trial is to investigate the effects of scapulothoracic exercises on postural stability, muscle strength, muscular endurance, mandibular functions and proprioception in sedentary individuals aged 18-45 years with head forward posture and temporomandibular joint dysfunction (Cranio-Cervico-Mandibular Malalignment). The main questions it aims to answer are:

• Do Scapulothoracic exercises given in addition to cervical posture exercises have an effect on postural stability, proprioception, muscle strength, muscular endurance and mandibular functions in individuals with Cranio-Cervico-Mandibular malalignment?

Researchers will compare conventional neck exercises (control group) and scapulothoracic exercises applied in addition to conventional neck exercises (treatment group) to see the effects of scapulothoracic exercises on the neck and jaw area.

DETAILED DESCRIPTION:
The investigators aimed to investigate the effects of scapulothoracic exercises on postural stability, muscle strength, muscular endurance, mandibular functions and proprioception in sedentary individuals aged 18-45 years with cranio-cervico-mandibular malalignment including head-first posture and temporomandibular joint dysfunction problems.

ELIGIBILITY:
Inclusion Criteria:

* Male and female students and employees between the ages of 18-45,
* Individuals with a craniovertabral angle (CVA) <50° and a Fonseca questionnaire score between 20-100,
* Individuals with a Helkimo clinical dysfunction index score between 1-25,
* Individuals with a low level of physical activity according to the International Physical Activity Questionnaire.

Exclusion Criteria:

* Serious problems of the musculoskeletal system, including the cervical and thoracic spine,
* Presence of serious chronic diseases such as hypertension, diabetes, cancer,
* Presence of neurological disease at a level that will affect balance and postural control,
* Being pregnant,
* Tooth and jaw problems in the last 6 months,
* Individuals with a total denture or prosthesis on the anterior teeth.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Postural Stability | Postural stability was measured at 3 different times (before treatment, 8 weeks after treatment, 12 weeks follow up). The average measurement time for each participant was 5 min.
  Five different data were obtained: the peripheral length value of the total sway degree (°) made on the device during balance, the percentile value of the area gap (%) showing the percentage of the area drawn according to the reference circle, the sway velocity value (°/sec), the average values (°) reached in the sway in the antero-posterior (AP) and medio-lateral (ML) directions.
Joint Position Sense | Proprioception measurements were made at 3 different times (before treatment, 8 weeks after treatment, 12 weeks follow up). The mean measurement time for mandibular position sense for each participant was 8 min. Cervical joint position sense measure
  Mandibular and cervical joint position sense measurements were made.

SECONDARY OUTCOMES:
Muscle Strength | Muscle strength measurements were made at 3 different times (pre-treatment, 8th week post-treatment, 12th-week follow-up). The temporomandibular joint depressor muscle strength measurement time for each participant lasted 3 minutes. The st
  Isometric muscle strength test will be performed on TMJ depressor muscles and cervical region muscles.
Endurance Measurement of Deep Neck Flexor Muscles | Muscular endurance of deep neck flexors was measured at 3 different times (pre-treatment, 8th week post-treatment, 12th week post-treatment follow-up). It took an average of 15 minutes for each participant.
  The muscular endurance measurement of the deep neck flexors will be made using the "craniocervical flexion test" and a stabilizer device.
Mandibular Function Disorder Questionnaire (MFBA) | Mandibular Function Disorder Questionnaire (MFBA) was measured at 3 different times (pre-treatment, 8th week post-treatment, 12th week post-treatment follow-up). It took an average of 2 minutes for each participant.
  It is used to evaluate the level of impairment in jaw functions in patients with TMED.

OTHER OUTCOMES:
Body Mass Index | Body Mass Index was measured at pre-treatment period.
  Height and body weights were measured to measure the body mass index of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Micoogullari, MSc, Principal Investigator — Cyprus International University
Locations (1):
- Cyprus International University, Mersin, Lefkosa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sajjadi, E., Olyaei, G. R., Talebian, S., Hadian, M. R., & Jalaie, S. (2014). The effect of forward head posture on cervical joint position sense. Archives of Advances in Biosciences, 5(4).
- [Background] Ryan, J., Akhter, R., Hassan, N., Hilton, G., Wickham, J., & Ibaragi, S. (2019). Epidemiology of temporomandibular disorder in the general population: A systematic review. Adv Dent Oral Health, 10(3), 1-13.
- [Background] Weber, P., Corrêa, E. C. R., de Paula Bolzan, G., dos Santos Ferreira, F., Soares, J. C., & da Silva, A. M. T. (2012). Relationship between craniocervical posture, mandible and hyoid bone and influence on alimentary functions. Brazilian Journal of Oral Sciences, 11(2), 141-147.
- [Background] Ries LG, Berzin F. Analysis of the postural stability in individuals with or without signs and symptoms of temporomandibular disorder. Braz Oral Res. 2008 Oct-Dec;22(4):378-83. doi: 10.1590/s1806-83242008000400016. PMID 19148396
- [Background] Gadotti I, Hicks K, Koscs E, Lynn B, Estrazulas J, Civitella F. Electromyography of the masticatory muscles during chewing in different head and neck postures - A pilot study. J Oral Biol Craniofac Res. 2020 Apr-Jun;10(2):23-27. doi: 10.1016/j.jobcr.2020.02.002. Epub 2020 Feb 5. PMID 32071851
- [Background] Moustafa IM, Youssef A, Ahbouch A, Tamim M, Harrison DE. Is forward head posture relevant to autonomic nervous system function and cervical sensorimotor control? Cross sectional study. Gait Posture. 2020 Mar;77:29-35. doi: 10.1016/j.gaitpost.2020.01.004. Epub 2020 Jan 7. PMID 31955048
- [Background] de Albuquerque Vieira, M., de Araújo, M. D. G. R., Antonino, G. B., da Silva Tenório, A., das Graças Paiva, M., & de Lima Ferreira, A. P. (2018). Cervical and scapular instability in subjects with temporomandibular disorder. Manual Therapy, Posturology & Rehabilitation Journal, 1-5.
- [Background] Chaves TC, Turci AM, Pinheiro CF, Sousa LM, Grossi DB. Static body postural misalignment in individuals with temporomandibular disorders: a systematic review. Braz J Phys Ther. 2014 Nov-Dec;18(6):481-501. doi: 10.1590/bjpt-rbf.2014.0061. Epub 2014 Oct 31. PMID 25590441
- [Background] Safwat͘, Y. M., Wadee, A. N., Lasheen, Y. R., & Kamel, R. M. (2019). Influence of Scapular Stabilization Exercises on Asymptomatic Forward Head Posture; A Randomized Controlled Trial. Indian Journal of Public Health Research & Development, 10(12).
- [Background] Dickerson SM, Weaver JM, Boyson AN, Thacker JA, Junak AA, Ritzline PD, Donaldson MB. The effectiveness of exercise therapy for temporomandibular dysfunction: a systematic review and meta-analysis. Clin Rehabil. 2017 Aug;31(8):1039-1048. doi: 10.1177/0269215516672275. Epub 2016 Oct 3. PMID 27697824
- [Background] Saito ET, Akashi PM, Sacco Ide C. Global body posture evaluation in patients with temporomandibular joint disorder. Clinics (Sao Paulo). 2009;64(1):35-9. doi: 10.1590/s1807-59322009000100007. PMID 19142549
- [Background] Zhao W, You H, Jiang S, Zhang H, Yang Y, Zhang M. Effect of Pro-kin visual feedback balance training system on gait stability in patients with cerebral small vessel disease. Medicine (Baltimore). 2019 Feb;98(7):e14503. doi: 10.1097/MD.0000000000014503. PMID 30762779